CLINICAL TRIAL: NCT05738148
Title: Vasopressin vs. Epinephrine During Neonatal Cardiopulmonary Resuscitation - a Cluster Randomized Controlled Phase I Trial
Brief Title: Vasopressin vs. Epinephrine During Neonatal Cardiopulmonary Resuscitation
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00122275
Record Dates: First submitted 2023-02-08; First posted 2023-02-21 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Cardiac Arrest Neonatal
MeSH Terms: interventions — Vasopressins; Epinephrine

STUDY DESIGN:
Intervention Model Description: Cluster-Crossover design
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Epinephrine (Active Comparator): Epinephrine group" Epinephrine will be administered according to current resuscitation guidelines either via umbilical vein catheter (0.02 mg/kg per dose) or via endotracheal tube (0.1 mg/kg) every three to five minutes as needed[2,3]. Chest compressions and epinephrine will be continued until ROSC.
  Interventions: Drug: Epinephrine
- Vasopressin (Experimental): "Vasopressin group" Vasopressin will be via umbilical vein catheter (0.4 IU/kg per dose - first line) or alternatively via an endotracheal tube (8 IU/kg) every three to five minutes as needed with a maximum of two doses if there is no ROSC [2,3] After that, the clinical team must convert to give epinephrine (0.02 mg/kg per dose) as long as CPR is ongoing.
  Interventions: Drug: Vasopressin

INTERVENTIONS:
Drug: Vasopressin — "Vasopressin group" Vasopressin will be via umbilical vein catheter (0.4 IU/kg per dose - first line) or alternatively via an endotracheal tube (8 IU/kg) every three to five minutes as needed with a maximum of two doses if there is no ROSC [2,3] After that, the clinical team must convert to give epinephrine (0.02 mg/kg per dose) as long as CPR is ongoing.
  Arms: Vasopressin
Drug: Epinephrine — "Epinephrine group" Epinephrine will be administered according to current resuscitation guidelines either via umbilical vein catheter (0.02 mg/kg per dose) or via endotracheal tube (0.1 mg/kg) every three to five minutes as needed[2,3]. Chest compressions and epinephrine will be continued until ROSC.
  Arms: Epinephrine

SUMMARY:
When a baby is born with a low heart rate or no heart rate, the clinical team must provide breathing support and chest compressions (what is call cardiopulmonary resuscitation or CPR). In some situations, the clinical team also need to give medications to help the heart rate increase. During CPR, the most common medication given is called epinephrine. There is another medication called vasopressin that is available that could be beneficial to newborn babies. However, no study has compared epinephrine with vasopressin in the delivery room during neonatal CPR.

The current study will be the first trial comparing this two medications during neonatal CPR.

The investigators will randomize our hospital to either epinephrine or vasopressin for the duration of one year. Babies will either receive CPR with epinephrine (this will be the control group) or CPR with vasopressin ( this will be the intervention group). The investigators believe that vasopressin may be more helpful to babies with a low heartrate or no heart rate at birth.

DETAILED DESCRIPTION:
Purpose

The infrequent need for CC and epinephrine during neonatal resuscitation, coupled with an inability to consistently anticipate which newborn infants are at high risk of requiring extensive CPR, explains the ongoing lack of high quality evidence (i.e., large randomized clinical trials) to better guide healthcare providers in their resuscitative effort. Guidelines for neonatal resuscitation recognized the lack of neonatal data and extrapolate data from studies with adults and adult/pediatric animal studies. Those data may not apply wholly to the neonatal population. Therefore, neonatal data are needed to determine the optimal vasopressor therapy during neonatal resuscitation.

Hypothesis

In newborns who require CPR does Vasopressin compared to Epinephrine reduce time to achieve return of spontaneous circulation defined as a heart rate of >60/min for 60sec .

Justification

Most newborn infants successfully make the transition from fetal to neonatal life without help. Between 10-20% of newborns (13-26 million worldwide) need respiratory support. In the delivery room, 0.1% of term infants and 10-15% of preterm infants (2-3 million worldwide) need cardiopulmonary resuscitation (CPR), defined as chest compressions (CC), 100% oxygen, and administration of the vasopressor drug, epinephrine. Despite receiving CPR, approximately 1 million of these newborns die every year worldwide. Newborn infants receiving extensive CPR in the delivery room have a high incidence of mortality (41%) and short-term neurologic morbidity (e.g., 57% hypoxic-ischemic encephalopathy and seizures). Further, newborns receiving epinephrine receiving epinephrine but with no signs of life at 10 minutes after birth had an 83% mortality rate and 93% of survivors will have moderate-to-severe disability. The poor prognosis associated with receiving epinephrine in the delivery room raises questions about whether using a specifically tailored vasopressor during neonatal CPR could improve outcomes.

Incidence of asphyxia in preterm and term newborns varies between 1-9/1000 and 1-2/1000 live births and represents the third most common cause of neonatal death. Asphyxia results from failure of placental gas exchange before delivery (e.g., abruption, chorioamnionitis) or deficient pulmonary gas exchange immediately after birth (e.g., apnea, respiratory distress syndrome). Asphyxia is impaired gas exchange with simultaneous hypoxia and hypercapnia. In >80% of asphyxiated neonates, it leads to mixed metabolic and respiratory acidosis plus dysfunction of one or more organ systems (including depressed myocardial function leading to cardiogenic shock, pulmonary hypertension, and ultimately cardiac arrest). The underlying etiology of bradycardia, and ultimately cardiac arrest, in neonates, results from severe hypoxemia, metabolic acidosis, and vascular compromise. This contrasts with the etiology most in adults, where onset of arrhythmias is followed by abrupt cessation of cardiac output in the setting of well-oxygenated blood. Ventilation is therefore more likely to be beneficial in neonatal CPR than in adult CPR.

In the asphyxiated and severely acidotic newborn, the vascular bed is maximally vasodilated with very low systemic vascular resistance. Providing CC will serve to mechanically pump the blood through the body until the myocardium becomes sufficiently oxygenated to maintain adequate output. Optimized CC can generate ~30% of normal organ perfusion, with preferential (>50%) perfusion to the heart and brain. The administration of systemic vasoconstrictors (epinephrine) induces intense peripheral vasoconstriction resulting in elevated systemic vascular resistance, enhanced diastolic blood flow, and increased coronary perfusion pressure (CPP) to improve coronary blood flow. However, in severely acidotic hemodynamically compromised lambs' intravenous epinephrine administration at 0.01 mg/kg did not improve cardiac output, heart rate or blood pressures.

Current neonatal resuscitation guidelines recommend administration of epinephrine once CPR has started at a dose of 0.02mg/kg preferably given intravenously (i.v.), with repeated doses every 3 min until ROSC. These recommendations are based on adult animal data, because neonatal data are lacking.

Epinephrine, is an endogenous catecholamine with high affinity for α1, α2, β1, and β2-receptors present in cardiac and vascular smooth muscle. Epinephrine causes vasoconstriction via stimulation of α1-receptors present in vascular smooth muscle, stimulation of α2-receptors causes presynaptic inhibition of norepinephrine release in the central nervous system and coronary vasoconstriction. Through β1-receptors, epinephrine increases heart rate (chronotropy), conduction velocity (dromotropy), contractility (inotropy), and rate of myocardial relaxation (lusitropy). β2-receptor stimulation leads to smooth muscle relaxation and in the myocardium increases contractility. However, epinephrine also increases myocardial oxygen demand and respiratory and metabolic acidosis, a common occurrence during neonatal asphyxia, and inhibits hemodynamic responses (e.g., aggravated hypertension, or tachycardia after ROSC). Furthermore in vivo effects of epinephrine depend on the i) dose of epinephrine, ii) number of receptors available on target tissues, iii) affinity of these receptors, and iv) local target tissue environments. Neonatal animal studies reported that 85% of asphyxiated piglets with cardiac arrest will require vasopressors to achieve ROSC[24,31-34]. There are some methodological flaws in these studies including i) these studies examined CC and reported vasopressor use as secondary outcomes only, ii) used a sheep model, which is not an ideal model, and iii) used the same dose in all studies. In addition, Sobotka et al reported that epinephrine administration (0.01 mg/kg) was a prerequisite for achieving ROSC, which occurred between 7-124sec after epinephrine administration in a transitional near-term lamb model of asphyxia-induced bradycardia. CC alone does not generate a sufficient diastolic blood pressure (a proxy for coronary artery perfusion pressure) to achieve ROSC[18]. Similarly, dp/dt (an assessment of diastolic function during isovolumic relaxation) only increases after epinephrine administration (0.02 mg/kg) compared to CC alone, which is associated with an increase in diastolic function, hence improved coronary artery perfusion pressure, which is a pre-requirement for ROSC. Similarly, Halling et al reported that 24/30 newborn infants required an average of 3 doses of epinephrine to achieve ROSC.

Alternatively, vasopressin, an antidiuretic hormone with vasoactive action through V1 receptor activation, is beneficial due to its postulated effects including combined pulmonary vasodilation and systemic vasoconstriction, not affected by respiratory and metabolic acidosis, and no increase in myocardial oxygen demand. Currently, a single dose of vasopressin at 40 international units (IU) is recommend during adult CPR, which is supported by several randomized trials[40]. Evidence from large randomized trials in adults reported that vasopressin is superior to epinephrine when cardiac arrest was caused by primary asystole. Wenzel et al compared vasopressin and epinephrine during out-of-hospital cardiac arrest in adults and reported similar rates of hospital admission in patients with ventricular fibrillation (46% vs. 43%) or pulseless electrical activity (34% vs. 31%). However, among patients with asystole, vasopressin was associated with significantly higher rates of hospital admission (29% vs. 20% p=0.02) and hospital discharge (5% vs. 2%, p=0.04). This suggests that vasopressin might be beneficial when asystole is the leading cause for cardiac arrest, when compared to that due to ventricular fibrillation or PEA.

Vasopressin may therefore be beneficial during neonatal CPR because in newborn infants i) asphyxia results primarily in non-shockable rhythm (asphyxia (40-45%) or pulseless electrical activity (40-50%), rather than ventricular fibrillation <5%).

Further, pulmonary vascular resistance is characteristically more prominent in newborns. Vasopressin's combined properties as pulmonary vasodilator and systemic vasoconstrictor properties of vasopressin might make it an ideal support drug in this context. However, evidence is limited on vasopressin effectiveness in pediatric or neonatal patients. Duncan et al reported that only 5% of the 1293 pediatric patients received vasopressin during in-hospital cardiac arrest. Although. patients who received vasopressin had a significantly longer duration of cardiac arrest (median 37 vs. 24min, p=0.004) and a longer time to ROSC, their survival at 24 hours or at discharge was similar to patients receiving epinephrine. A recent feasibility study compared vasopressin (0.8IU/kg) after an initial epinephrine dose in patients <18 years of age (n=10) to ≥ two doses of epinephrine. Patients who received vasopressin had increased 24-hr survival (80% vs. 30%, odds ratio (OR) (95%CI) 9.3 (1.5-57.7)), with similar time to ROSC, survival to hospital discharge, and neurologic status at discharge. Until now only one study has compared vasopressin with epinephrine in a neonatal piglet model of cardiac arrest. The study reported higher survival rates with vasopressin vs. epinephrine [16/20 vs. 11/24 (p<0.05)] with less myocardial necrosis on autopsy.

Both asphyxiated piglets and newborn infants require epinephrine to achieve ROSC. Further, there is only a 20% success rate after a single dose of i.v. epinephrine, with multiple doses needed by many newborns. During asphyxiated in pediatric patients (~6 years of age) there was no improvement in ROSC but increased mortality after epinephrine administration. Thus, an alternative vasopressors therapy might improve outcomes. In adult patients, vasopressin compared to epinephrine was associated with increased rates of ROSC [OR (95% CI) 1.70 (1.17, 2.47), p=0.005] and higher long-term survival [OR (95% CI) 1.80 (1.04, 3.12), p=0.04. Therefore, vasopressin might reduce time to ROSC and improve outcomes for asphyxiated newborn infants. While there are several animal and neonatal cohort studies examining epinephrine, studies examined vasopressin are lacking.

The investigators compared vasopressin and epinephrine in our established piglet model of neonatal asphyxia and observed that mean (SD) time to ROSC with epinephrine (0.02 mg/kg with 342 (194)sec, respectively, compared vasopressin (0.2, 0.4, and 0.8 IU/kg with 115(35) 149(86), and 121(44)sec), respectively.

Furthermore, cardiovascular parameters including heart rate, carotid blood flow, mean arterial pressure (MAP), cerebral oxygenation (Brain SO2) were also improved with Vasopressin, most effectively with 0.4, IU/kg.

Alternative administration of vasopressin endotracheal compared to epinephrine resulted in increases of up to 180% in diastolic blood pressure and up to 140% in systolic blood pressure, which are both essential for successful resuscitation.

These data suggest, that clinical data are needed to assess if vasopressin might be an alternative for epinephrine.

ELIGIBILITY:
Inclusion criteria Infants (term or preterm infants) born without heart beat or with bradycardia

Exclusion criteria:

Congenital heart disease (e.g., hypo-plastic left heart) Condition that have adverse effect on breathing or ventilation (e.g., congenital diaphragmatic hernia), o

Ages: 0 Minutes to 20 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2026-01-13 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Time to ROSC (Return of spontaneous Circulation) | up to 60 Minutes of chest compression
  Duration of Chest Compression until heart rate increases to greater 60 beats per minute, which is maintained for 60sec.

SECONDARY OUTCOMES:
Mortality | Within the first 28 days
  Number of infants who die until discharge - comparison between group
Number of Patients who have brain injury | Until infant is discharge from hospital (maximum of 30 weeks after birth)
  Brain injury either by ultrasound or magnet resonance imaging - comparison between group
Number of Epinephrine doses during resuscitation | During resuscitation (up to 60 minutes)
  How many doses of epinephrine are given
Number of Vasopressin doses during resuscitation | During resuscitation (up to 60 minutes)
  How many doses of epinephrine are given
Admission temperature | within 60 minutes after birth
  body temperature at admission after birth
Use of therapeutic cooling | First 72 hours after birth
  Number of infants who receive therapeutic cooling during hospital admission
Mode of mechanical ventilation | Until infant is discharge from hospital (maximum of 30 weeks after birth)
  Number of infants who receive mechanical ventilation during hospital admission
Cerebral regional oxygen saturation | First 72 hours after birth
  Changes in Cerebral regional oxygen saturation measured using near-infrared spectrocopy
Mask ventilation in the delivery room | up to 60 Minutes
  Number of infants who receive mask ventilation during chest compression
Intubation in the delivery room | up to 60 Minutes
  Number of infants who were intubated during chest compression
Acute Kidney injury | 24 hours after birth
  To assess serum creatinine and cumulative urine output
Blood gases and serum sodium levels | 8-12 hours after birth
  To assess blood gas values (i.e., pH, paCO2, Base excess) and Sodium blood concertation
Blood gases and serum sodium levels | 24-28 hours after birth
  To assess blood gas values (i.e., pH, paCO2, Base excess) and Sodium blood concertation

CONTACTS AND LOCATIONS:
Overall Officials: Georg Schmolzer, Principal Investigator — University of Alberta
Locations (1):
- Royal Alexandra Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
The trial dataset will be stored and maintained at the Royal Alexandra Hospital, where it will be accessible to all trial investigators for quality monitoring.
  Other access to the study data will be available by request to the principal investigator.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: study protocol and ICF are available upon request, SAP and analytic code in 2027
Access Criteria: Data requestors seeking to use trial data to generate new publications or presentations will be asked to submit a proposal that will be reviewed by the principal investigator and co-investigators.

REFERENCES:
- [Derived] Ramsie M, Cheung PY, Law B, Schmolzer GM. Vasopressin versus epinephrine during cardiopulmonary resuscitation of asphyxiated newborns: A study protocol for a prospective, cluster, open label, single-center, randomized controlled phase 2 trial - The VERSE-Trial. Resusc Plus. 2023 Aug 31;16:100459. doi: 10.1016/j.resplu.2023.100459. eCollection 2023 Dec. PMID 37663146